CLINICAL TRIAL: NCT00512837
Title: A Mobile Phone Based Structured Intervention to Achieve Asthma Control in Patients With Uncontrolled Persistent Asthma: Pragmatic Randomised Controlled Trial
Brief Title: Mobile Phone Based Structured Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 07/047
Record Dates: First submitted 2007-08-07; First posted 2007-08-08 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2008-06

CONDITIONS: Asthma
Keywords: Telemedicine; clinical management; empowerment; engagement; education
MeSH Terms: conditions — Asthma; Empowerment

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 2 (Active Comparator)
  Interventions: Behavioral: Mobile phone technology

INTERVENTIONS:
Behavioral: Mobile phone technology

SUMMARY:
Although asthma outcomes can be improved with structured care, less than half of people with asthma achieve good control. Part of the problem is poor adherence with self-monitoring and preventive drug regimes. This trial will test whether using mobile phone-based monitoring, as part of a structured care plan, improves clinical outcomes and confidence in people with poorly controlled asthma.

Adults and teenagers with poorly controlled asthma will be recruited and randomly assigned to one of two groups. Those in the mobile phone group will monitor their asthma daily using their mobile phone to record symptoms, medication and lung function. Instantaneous feedback to their phone will provide a visual indication of asthma control and prompts about therapy. The patient and their clinician will have web-based access to all readings. People in the control group will use traditional paper-based monitoring. Under the care of their asthma nurse, both groups will be treated according to the step-wise approach of the BTS/SIGN asthma guideline in order to gain control.

We will use the validated Asthma Control Questionnaire to measure control at baseline, three and six months, and compare improvement in the two groups. We will also assess how confident people feel in controlling their asthma, using a validated measure of self-efficacy, attitudes and knowledge.

Technological solutions to long-term healthcare problems are increasingly being sought by patients, clinicians and policy makers. If successful, our trial could provide timely evidence for the use of information technology to address the long-recognised problem of poor asthma control.

DETAILED DESCRIPTION:
A. Hypothesis In teenagers and adults with poorly controlled asthma offered treatment according to BTS-SIGN guideline, the use of mobile phone-based lung function and symptom monitoring with patient feedback will improve the asthma control achieved and patient self-efficacy at six-months compared to usual paper-based monitoring strategies.

B. Background Despite effective treatments, studies continue to demonstrate that asthma is poorly controlled,1,2 though marked variation in the control achieved in UK general practices suggests that improvement is possible for the vast majority of patients.3 Psychosocial factors such as denial of illness, low outcome expectations 4,5 and hectic lifestyles, exacerbated by limited knowledge, poor self-recognition of symptoms and discordant attitudes, influence patients' ability to engage in self-management with resultant poor concordance with monitoring and treatment.6,7 Interventions involving biofeedback can address these barriers by objectively demonstrating symptom severity and the impact of medication compliance.8 A Cochrane review demonstrates that self-management education linked with structured care improves asthma outcomes.9 Despite self-management education,6 in real life, compliance with traditional diary monitoring can be as low as 6%,10 and results are often fabricated.11 Electronic recording may improve compliance,12 with over two-thirds of potential readings recorded over a 72-week trial.13 Increasingly pervasive throughout society, mobile phone technology provides a convenient, portable communications medium. Mobile phone-based monitoring with supporting biofeedback, appears able to engage patients in their management, resulting in high levels of adherence and patient acceptability,13,14 with many patients welcoming the innovative care.15,16,17,18 Integrated within a structured care protocol, this has the potential to address the barriers of poor adherence and low expectations and thereby to improve patient outcomes.

Monitoring is, in itself, an intervention which alters behaviour. The theoretical model developed by Glasziou et al. describes the complementary and evolving roles of periodic professional reviews and on-going patient self-monitoring.19 The monitoring of asthma with lung function and/or symptoms is cited as a well-defined exemplar of this concept. Our recent qualitative study suggests that people with asthma perceive a role for mobile technology in aiding transition from clinician-supported phases while control is gained, to effective self-management during maintenance phases.20 This approach resonates with two key health service policies: the drive for technological solutions to healthcare problems;21 and the importance of expert patients and self-management of long-term conditions.22,23 Our proposed trial tests the hypothesis that through engaging the patient in self-monitoring with timely biofeedback, mobile phone technology can improve the asthma control achieved at six months compared to usual paper-based monitoring.

Our multi-disciplinary team has extensive experience of tele-care, delivery of primary care respiratory services, patient self-management, and research within general practice settings. Building on extensive background work,3,13-15,17,18,20 we offer expertise in respiratory and health services research, and social science and are ideally placed to undertake this trial.

Description of the mobile phone-based monitoring system (see figure) The system software (T+ asthma, Oxford, UK) can be loaded onto any web-enabled mobile phone. It permits recording of symptoms, medication usage and lung function. Measurements are made with a Piko meter (a prescribable electronic meter which records both (FEV1) and peak expiratory flow (PEF)). We have opted to record FEV1 because it is a component of the ACQ,24 and the correlation between Piko and spirometry FEV1 is excellent (r=0.98).25,26 Data transmitted to a remote server are analysed and the latest reading returned to the mobile phone, compared with the preceding week's recordings and a prompt for using 'preventer' medication. In addition, the patient and their clinician can access the record via a password-protected website.C. Design of the research A six month single-blinded randomised controlled trial

Practice recruitment Six/eight practices (total list 72,000 patients) will be recruited from the Leicester area (local to the practice of a lead co-applicant). Eligible practices will have an asthma-trained nurse able to commit to the additional clinical workload.

Participant recruitment Practices will use the Minimal Asthma Assessment Tool (MAAT), which interrogates routinely collected data on their computer database, using patterns of medication usage, symptom control and biometric data to identify patients (12 years and over) with poorly controlled asthma.3 Potential eligibility will be confirmed by inspection of manual/computer records checking (and documenting) exclusion criteria: other significant lung disease, under specialist care for severe/difficult asthma, unable to communicate in English or use a mobile phone and at the request of the GP for other significant social/clinical problems. The practice will invite all potentially eligible patients by post to participate.

Confirmation of eligibility and baseline assessment Potential participants will attend a screening assessment (normally in their practice) at which eligibility will be confirmed, their current asthma control assessed using the ACQ,24 and suitability of their mobile phone established. All patients with poorly controlled asthma (defined as ACQ>1.5 27) will be entered in the trial and a baseline assessment undertaken.(see summary table)

Randomisation Patients will be allocated, using centralised randomisation stratified by practice, to mobile phone or paper-based monitoring. The University of Aberdeen's Health Services Research Unit will provide a 24hr telephone randomisation service.

Intervention group: Mobile phone based monitoring Patients in the intervention group will be issued with a Piko meter and the T+ software loaded onto their mobile phone. They will be asked to monitor symptoms, medication usage and FEV1 twice a day and submit the readings. The web-record will be available to patient and asthma nurse to aid assessment of control during routine reviews, and to the patients' GP in the event of unscheduled asthma consultations.

Control group: paper-based monitoring Patients in the control group will be issued with a Piko meter, and asked to keep a paper diary, recording symptoms, medication usage and FEV1 readings twice a day.

Clinical care and self-management education in both groups Structured care will be provided by the practices' asthma nurse(s), trained in all aspects of the trial.

Clinical care in both groups will be in accordance with the step-wise approach of the BTS-SIGN Guideline.28 Patients will be reviewed monthly until control is achieved as judged by the nurse on the basis of clinical monitoring.

All patients will receive a one-to-one standardised asthma education session, including information on asthma, asthma treatment, inhaler technique, monitoring and when to seek urgent assistance.

ELIGIBILITY:
Inclusion Criteria:

* Patient with poorly controlled asthma

Exclusion Criteria:

* Patient under age of 12
* Not possessing a mobile phone and who don't have adequate command of the English language

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
change in asthma control between baseline and six months as measured by ACQ.24 The ACQ measures clinical goals of asthma management on a scale: 0 (good control) to 6, is responsive to change,24 with a intra-individual minimum important difference | 6 months

SECONDARY OUTCOMES:
Morbidity • Mean difference in ACQ at 3 and 6 months.24,36 • Proportion of patients with an ACQ<0.75 at three and six months.27 • Mean difference in mini-AQLQ which measures the physical/emotional impact of asthma on a scale

CONTACTS AND LOCATIONS:
Overall Officials: Dermot Ryan, Principal Investigator — Univeristy of Aberdeen
Locations (1):
- Dr Jones and Partner, Norfolk, United Kingdom

REFERENCES:
- [Derived] Cox NS, Dal Corso S, Hansen H, McDonald CF, Hill CJ, Zanaboni P, Alison JA, O'Halloran P, Macdonald H, Holland AE. Telerehabilitation for chronic respiratory disease. Cochrane Database Syst Rev. 2021 Jan 29;1(1):CD013040. doi: 10.1002/14651858.CD013040.pub2. PMID 33511633
- [Derived] Ryan D, Price D, Musgrave SD, Malhotra S, Lee AJ, Ayansina D, Sheikh A, Tarassenko L, Pagliari C, Pinnock H. Clinical and cost effectiveness of mobile phone supported self monitoring of asthma: multicentre randomised controlled trial. BMJ. 2012 Mar 23;344:e1756. doi: 10.1136/bmj.e1756. PMID 22446569
- [Derived] Ryan D, Pinnock H, Lee AJ, Tarassenko L, Pagliari C, Sheikh A, Price D. The CYMPLA trial. Mobile phone-based structured intervention to achieve asthma control in patients with uncontrolled persistent asthma: a pragmatic randomised controlled trial. Prim Care Respir J. 2009 Dec;18(4):343-5. doi: 10.4104/pcrj.2009.00064. No abstract available. PMID 19940961